CLINICAL TRIAL: NCT02761720
Title: Mobile App for Mood in Pregnancy (Ginger iO)
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Ginger.io (Industry)
Responsible Party: Sponsor
Other Study IDs: 821784
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Mood Disorders; Depression
MeSH Terms: conditions — Mood Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- MyPennMedicine (MPM): Participants assigned to this arm downloaded only the MyPennMedicine mobile app.
  Interventions: Other: No Intervention
- MPM and Ginger iO: Participants assigned to this arm downloaded both the MyPennMedicine mobile app and Ginger iO mood tracking app.
  Interventions: Other: No Intervention
- Lottery: Participants assigned to this arm downloaded both the MyPennMedicine mobile app and Ginger iO mood tracking app. They were also given a lottery incentive if they completed 70% of the daily mood ratings.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The Mobile Mood Tracking App study is a small randomized trial of acceptability and usability of a mobile phone mood tracking application (mobile app) among women with depressed mood in pregnancy. The study will be assessing the perceived value and usability of this tool in pregnancy over eight weeks to test whether women using this app are more likely to receive assessments and treatments of depressed mood than women not using it.

ELIGIBILITY:
Inclusion Criteria:

* Positive screening for elevated depression symptomatology (PHQ-9 score must be greater than or equal to 5.)

Exclusion Criteria:

* Women with pregnancies of less than 33 weeks gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Dickens Center provides prenatal care to women with Medicaid insurance and its predominantly African American (90%). The mean age of patients receiving prenatal care is 25 years in this site.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evidence of increased provider intervention for the treatment of worsening depressive symptoms confirmed by the mobile mood tracking application. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dickens Center for Women's Health at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States